CLINICAL TRIAL: NCT05066750
Title: What Makes People Better at Retrieving Difficult Words?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Colorado Springs (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Lori James, Professor, University of Colorado, Colorado Springs
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2020-005; R15AG063111-01 (NIH)
Record Dates: First submitted 2021-09-08; First posted 2021-10-04 (Actual); Results first posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Healthy Aging
Keywords: mindful breathing; anxiety; word retrieval
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of two behavioral intervention conditions before performing a word retrieval task
Who Masked: Participant
Masking Description: Participants in each condition do not know what other participants are doing, nor that there is another condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindful breathing video (Experimental): Participants watch a 10 minute mindful breathing video
  Interventions: Behavioral: Mindful breathing
- Control video (Active Comparator): Participants watch a 10 minute control video
  Interventions: Behavioral: Control video

INTERVENTIONS:
Behavioral: Mindful breathing — Participants watch a 10 minute mindful breathing video
  Arms: Mindful breathing video
Behavioral: Control video — Participants watch a 10 minute control video
  Arms: Control video

SUMMARY:
This study is being conducted to learn more about how various personal and situational characteristics are related to the ability to produce words in response to definitions. Participants will watch a video, then see definitions and try to come up with a word that fits each one. Participants will also complete some surveys and other measures. Collected data will give researchers a better understanding of how individuals' personality and cognitive traits and setting in which word retrieval occurs relate to the ability to produce individual words.

DETAILED DESCRIPTION:
This study is being conducted to learn more about how various personal and situational characteristics are related to the ability to produce words in response to definitions. Adult participants ages 18-30 and 65-80 will participate in videoconference calls during which a video is shown and definitions are presented. Participants will try to come up with a word that fits each definition, and then complete some surveys, including some about anxiety, mindfulness, attention, vocabulary, and demographics. Participation will take approximately 1.25 hours. Collected data will be de-identified, and the aggregate data will give researchers a better understanding of how individuals' personality and cognitive traits and setting in which word retrieval occurs relate to peoples' ability to produce individual words.

ELIGIBILITY:
Inclusion Criteria:

* fluent speakers of English ages 18-30 or ages 65-80

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2021-08-23 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2022-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lori James, PhD, Principal Investigator — University of Colorado, Colorado Springs
Locations (1):
- UCCS, Colorado Springs, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
De-identified participant data may be posted on a website for open access to other researchers, if the publication outlet requires it, but it is not currently planned.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mindful Breathing Video | Control Video
Started | 85 | 85
Analysis Population | 85 | 83
Completed | 85 | 85
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mindful Breathing Video | Control Video | Total
Number analyzed (Participants) | 85 | 85 | 170
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 42 | 43 | 85
  >=65 years | 43 | 42 | 85
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 62 | 120
  Male | 27 | 23 | 50
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 74 | 71 | 145
  More than one race | 6 | 9 | 15
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 85 | 85 | 170

OUTCOME MEASURES:

1. Primary Outcome: Word Retrieval Performance
Description: Percent of trials with correct responses and percent of trials that are word retrieval failures will be measured on a task created for this purpose. Specifically, participants will try to provide words that best fit definitions, indicating when a word gets stuck on the "tip of their tongue."
Time Frame: During the 1.25 hour experimental session
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Mindful Breathing Video | Control Video
Number analyzed (Participants) | 85 | 83
Percent
  Percent correct | 41 (19) | 37 (18)
  Percent TOTs | 11 (7) | 11 (7)

ADVERSE EVENTS:
Time Frame: During 1.25 hour experimental session
Description: This is a minimal risk experiment so no risk of adverse events beyond everyday life
Arm/Group | Mindful Breathing Video | Control Video
All-Cause Mortality (participants affected / at risk) | 0/85 | 0/85
Serious Adverse Events (participants affected / at risk) | 0/85 | 0/85
Other Adverse Events (participants affected / at risk) | 0/85 | 0/85

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-02-11): https://cdn.clinicaltrials.gov/large-docs/50/NCT05066750/Prot_000.pdf
  • Informed Consent Form (2022-01-03): https://cdn.clinicaltrials.gov/large-docs/50/NCT05066750/ICF_001.pdf